CLINICAL TRIAL: NCT05231993
Title: Clinical Triage and Treatment of Atypical Glandular Cells (AGC) Detected in Screening: Randomized Healthservices Trial
Brief Title: Clinical Triage and Treatment of Atypical Glandular Cells (AGC) Detected in Screening
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Regional Cancer Centre Stockholm Gotland (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Joakim Dillner, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AGC
Record Dates: First submitted 2022-01-29; First posted 2022-02-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Uterine Cervical Cancer
Keywords: cervical cancer, atypical glandular cells
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Conization; Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active comparator (Active Comparator): 1. All women ages <41, women ages ≥41 with TZ1 and TZ2, and women ages ≥41 with a desire for further childbearing Clinical management and follow-up according to the national screening guidelines published in 2017 (same as for the comparator group, see below).
  2. Women with TZ3 and women ages ≥41 with no desire for further childbearing a. Referral to (diagnostic) excision. The depth of the diagnostic excision will be clinically determined in the trial. It should be with the intent to treat but no so extensive that the risk for side effects increases.
  The excision should include a cervical abrasion and endometrial sampling.
  Interventions: Procedure: Conization
- Placebo comparator (Placebo Comparator): Clinical management and follow-up according to the national screening guidelines published in 2017:
  1. Colposcopy with biopsy within 3 months, endocervical sample, ultrasound and endometrial biopsy if the woman is ≥40
  2. Colposcopy after 12 months if the first colposcopy and biopsies are normal
  3. Cytology and HPV testing at 12 and 24 months if the second colposcopy is normal
  Interventions: Procedure: Colposcopy

INTERVENTIONS:
Procedure: Conization — A cone biopsy to remove abnormal tissue.
  Other Names: Excision
  Arms: Active comparator
Procedure: Colposcopy — 1. Colposcopy with biopsy within 3 months,endocervical sample, ultrasound and endometrial biopsy if the woman is ≥40
  2. Colposcopy after 12 months if the first colposcopy and biopsies are normal
  3. Cytology and HPV testing at 12 and 24 months if the second colposcopy is normal
  Arms: Placebo comparator

SUMMARY:
The risk of cervical cancer after diagnosis with atypical glandular cells (AGC) detected by screening is elevated for 15 years after discovery. The current recommendation is that when AGC is detected during screening, referel is made to a gynecologist for colposcopy with biopsy within 3 months after the index test. Repeated tests should be done after one year and after two years and if these are negative, the woman can return to routine screening.

Given the increased risk of cancer associated with AGC a new evaluation of the optimal follow-up and treatment of AGC, which is detected during screening, is carried out. In this randomized study, women with AGC will be randomized to routine treatment according to current guidelines or to conization. The aim of the study is to determine which of the two treatments is most effective.

DETAILED DESCRIPTION:
Evidence from a nationwide cohort study demonstrated that the risk of cervical cancer following a diagnosis of AGC detected in screening was elevated for 15 years, particularly the risk of adenocarcinoma. Furthermore, the study suggested that compared to high-grade squamous intraepithelial lesion (HSIL) management, the management of AGC has been suboptimal in Sweden (Wang et al., BMJ 2016). A study conducted in the greater metropolitan region of Stockholm showed that the PPV for high grade lesions was 60% for Human Papillomavirus (HPV) positive AGC detected in screening (Norman et al., BMJ Open, 2017).

The new guidelines for cervical cancer prevention were adopted in January of 2017 nationally and in December 2017 in county of Stockholm and outline a clinical management strategy for AGC. The recommendation is that AGC detected in screening, regardless of HPV status, should be referred to a gynecologist for colposcopy with biopsy within 3 months of the index test. For women over the age of 40, an ultrasound and endometrial biopsy is also recommended. Repeat tests should be done at one year and two years, if these are negative then the woman can return to routine screening.

The elevated risk for high grade lesions and cancer associated with AGC, coupled with the reality that cervical cancer incidence has increased in Sweden, begs a new evaluation of the optimal clinical management and treatment of AGC detected in screening. Women will be randomized to routine management according to the new guidelines or to an alternative management.

ELIGIBILITY:
Inclusion Criteria:

* give informed consent
* Women diagnosed with AGC (atypical glandular cells, M69720) and HPV 16/18 positive, detected in cervical screening.

Exclusion Criteria:

* Do not give informed consent
* HPV negative or none-HPV16/18 positive

Ages: 23 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
CIN3+ | 2-3 years
  Proportion of women with histologically verified HSIL+ (CIN3+) including AIS+ after AGC found in screening

SECONDARY OUTCOMES:
CIN2+ | 2-3 years
  Proportion of women with histologically verified HSIL+ (CIN2+) including AIS+ after AGC found in screening

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Elfgren, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
To be determined.

REFERENCES:
- [Result] Norman I, Hjerpe A, Dillner J. Risk of high-grade lesions after atypical glandular cells in cervical screening: a population-based cohort study. BMJ Open. 2017 Dec 14;7(12):e017070. doi: 10.1136/bmjopen-2017-017070. PMID 29247086
- [Result] Wang J, Andrae B, Sundstrom K, Strom P, Ploner A, Elfstrom KM, Arnheim-Dahlstrom L, Dillner J, Sparen P. Risk of invasive cervical cancer after atypical glandular cells in cervical screening: nationwide cohort study. BMJ. 2016 Feb 11;352:i276. doi: 10.1136/bmj.i276. PMID 26869597